CLINICAL TRIAL: NCT05195801
Title: Intraoperative Optic Nerve Diameter and Intraocular Pressure Changes in Patients Undergoing Vitrectomy (PPV) Surgery Under General Anesthesia and Their Effects on Vision in the Postoperative Period
Brief Title: Optic Nerve Diameter and Intraocular Pressure Changes in Patients Undergoing Vitrectomy Under General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, İlker Onguc Aycan, Professor, MD, Akdeniz University
Other Study IDs: Effect of GA on vision in PPV
Record Dates: First submitted 2022-01-07; First posted 2022-01-19 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Vision Disorders; Ocular Surface Disease
Keywords: vitrectomy; general anaesthesia; optic nerve; intraocular pressure; vision field
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group with local anesthesia: The group that did not apply general anesthesia
  Interventions: Device: USG
- Group with Sevoflurane: The Sevoflurane used for maintenance of general anesthesia
  Interventions: Device: USG
- Group with Propofol: The Propofol (IV) used for maintenance of general anesthesia
  Interventions: Device: USG

INTERVENTIONS:
Device: USG — Optic Nerve Diameter will be measured in the intraoperative period and postoperative 1st month by ultrasonography method.

SUMMARY:
This study aimed to measure optic nerve sheath changes in the intraoperative period in patients who underwent vitrectomy surgery and to investigate the intraoperative factors that may affect this.

Standard anesthesia protocol will be applied to all patients participating in the study. Optic nerve sheath diameter measurements of the patients taken to the operating room will be made on the operating table by ultrasonography method. Standard anesthesia induction will be performed following SpO2 and ECG monitoring in routine anesthesia monitoring. Depth of anesthesia will be evaluated with routine hemodynamic data.

DETAILED DESCRIPTION:
The optic nerve is part of the central nervous system and is surrounded by the dura, arachnoid, and pia mater; The sheath surrounding the optic nerve is in continuity with the dura mater of the brain and the subarachnoidal space filled with cerebrospinal fluid (CSF), creating a direct connection between the two chambers. (1) The optic nerve sheath continues the dura mater, and the subarachnoid space contains CSF. Thus, any increase in ICP in the subarachnoid space is transferred to the fluid in the optic nerve surrounding it. Because the optic nerve (ONS) can expand, changes in CSF pressure affect the volume of the optic nerve diameter (ONSD) with fluctuations in the anterior retrobulbar compartment, about 3 mm behind the globe. ONSD measurement for CT, MRI, and ultrasound-based intracranial pressure (ICP) detection has been studied previously. Ultrasonography has the potential advantage of being a reproducible, safe, and low-cost tool at the bedside without the risk of radiation and side effects. Sonographic ONSD measurement is made using a linear probe that is carefully placed on the closed upper eyelid without applying pressure to the eye while the patient is in the supine position. (2) Recently, studies have reported that measuring optic nerve sheath diameter (ONSD) using non-invasive imaging technologies provides alternative markers for early rising ICP. (1,2) The retina is the innermost tissue layer of the back of the eye. It consists of multiple layers of cells. The outermost layer is adjacent to the vitreal space and the choroid's innermost layer. Retinal detachment is when the neurosensory retina loses its adhesion to the underlying retinal pigment epithelium (RPE). The outer part of the neurosensory retina is where the photoreceptors are located. The choroid provides oxygen and nutrients for the photoreceptors. There are no retinal blood vessels in the fovea, and the retinal tissue in this area is entirely dependent on the choroid for oxygen requirements. Detachment of the macula can cause permanent damage to the photoreceptors in this location. Vision can be preserved if the macula remains attached and the retina is reattached correctly. (3) There are three categories of retinal detachment: rhegmatogenous, tractional, and exudative. Ruptured retinal detachments are the most common and are caused by fluid passing from the vitreous cavity through a retinal tear or entering the potential space between the sensory retina and the RPE. Tractional detachments occur when the proliferative membranes contract and elevate the retina. Components of rhegmatogenous and tractional etiologies may also lead to retinal detachment. Exudative detachments are caused by fluid buildup under the sensory retina caused by retinal or choroidal diseases. (3) The treatment of torn and tractional retinal detachments is typically surgical. Exudative macular detachments usually have nonsurgical treatment. The prognosis of retinal detachment varies greatly depending on the type of detachment and patient presentation. One of the most important prognostic factors for retinal detachment is whether the macula remains attached. If the macula remains attached, the time until surgery does not change the final visual result. However, the visual prognosis is relatively poor if the macula is detached. (3) Anesthetic agents may affect the ICP during surgery. A dose-dependent decrease in cerebral blood flow, cerebral metabolic rate, and ICP have been reported with propofol anesthesia. Sevoflurane is a cerebral vasodilator that can increase cerebral blood flow, cerebral blood volume, and ICP in a dose-dependent manner. (4)

Anesthetics suppress the activity of the electroencephalogram and reduce the cerebral metabolic rate. However, changes in cerebral metabolic rate and cerebral blood flow are not constant and depend on how anesthesia affects cerebral vascular smooth muscle. Sevoflurane has a dose-dependent effect on vascular smooth muscle relaxation and intrinsic cerebral vasodilator activity through direct inhibition of several pathways. Therefore, cerebral blood flow increases significantly during sevoflurane anesthesia, and ICP may increase as a result. However, propofol slows down EEG activity, reduces adenosine consumption rate, and decreases cerebral metabolic rate. Decreased cerebral metabolic rate decreases cerebral blood flow and cerebral blood perfusion, which decreases ICP. In addition, previous human and animal studies have determined that propofol leads to a progressive decrease in ICP. (4) This study aimed to measure optic nerve sheath changes in the intraoperative period in patients who underwent vitrectomy surgery and to investigate the intraoperative factors that may affect this.

Standard anesthesia protocol will be applied to all patients participating in the study. Optic nerve sheath diameter measurements of the patients taken to the operating room will be made on the operating table by ultrasonography method. Standard anesthesia induction will be performed following SpO2 and ECG monitoring in routine anesthesia monitoring. Depth of anesthesia will be evaluated with routine hemodynamic data.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Taken to elective vitrectomy surgery
* Asa I - II - III patients
* GKS 15

Exclusion Criteria:

* Emergency surgeries
* Patients with a GCS of less than 15 or whose cognitive functions have not been evaluated as clinically sufficient.
* In cases that cause the termination of the surgical procedure for any reason during the operation
* Patients followed by neurosurgery and patients with intracranial events

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing vitrectomy surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Optic Nerve Diameter | one month
  This study aims to use the anesthesia methods routinely applied in our hospital's vitrectomy operations. With general anesthesia, intracranial pressure changes, an indication of which is an increase in the diameter of the optic nerve sheath. The expected benefit of this study is to reveal the effects of general anesthesia, patient profile (age, comorbidity, BMI), ventilator parameters on optic nerve sheath diameter in patients undergoing vitrectomy surgery, and to provide optimal intraoperative conditions in the surgery of these patients with parameters that can be corrected and to improve their vision in the postoperative period.
  The optic nerve diameter will be measured at determined time intervals, and changes in diameter will be noted in the study.

SECONDARY OUTCOMES:
Vision field | one month
  Changes in the patients' vision field will be measured in the postoperative period.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Akdeniz University Medical Faculty Department of Anesthesiology and Reanimation, Antalya
  - Akdeniz University Hospital, Antalya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen LM, Wang LJ, Hu Y, Jiang XH, Wang YZ, Xing YQ. Ultrasonic measurement of optic nerve sheath diameter: a non-invasive surrogate approach for dynamic, real-time evaluation of intracranial pressure. Br J Ophthalmol. 2019 Apr;103(4):437-441. doi: 10.1136/bjophthalmol-2018-312934. Epub 2018 Oct 25. PMID 30361274
- [Background] Robba C, Santori G, Czosnyka M, Corradi F, Bragazzi N, Padayachy L, Taccone FS, Citerio G. Optic nerve sheath diameter measured sonographically as non-invasive estimator of intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2018 Aug;44(8):1284-1294. doi: 10.1007/s00134-018-5305-7. Epub 2018 Jul 17. PMID 30019201
- [Background] Blair K, Czyz CN. Retinal Detachment. 2024 Feb 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK551502/ PMID 31855346
- [Background] Illarionov AM. [The blood coagulation and its fibrinolytic activity in patients who have sustained an apoplectic stroke]. Sov Med. 1966 Feb;29(2):76-7. No abstract available. Russian. PMID 6011519